CLINICAL TRIAL: NCT06812312
Title: Impact of Basic Cardiopulmonary Resuscitation on the Knowledge and Attitude of Professional Football Players and Coaches
Acronym: VILRCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Villarreal CF (Unknown); Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Isabel Almodóvar Fernández, Doctor, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Jugadores RCP
Record Dates: First submitted 2025-01-25; First posted 2025-02-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: CPR Skills; CPR Quality Assessment; CPR; Football Players; Coaches
Keywords: cardiopulmonary resuscitation; knowledge; attitude; nursing; professional soccer; Spain
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This study was conducted in two phases:
  The first phase consisted of an observational cross-sectional study with 206 participants who completed the questionnaires in person.
  The second phase consisted of an educational intervention with pre-post intra-subject control over 70 participants, conducted online.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention with pre-post intra-subject (Experimental): The sampling carried out was non-probabilistic and incidental. Inclusion criteria included being professional football players or coaches in the Valencian Community. A two-hour training intervention was conducted by a CPR-B instructor. The first 30 minutes were dedicated to explaining how to recognize a cardiopulmonary arrest, the correct technique for chest compressions, ventilations, and AED use. The remaining 90 minutes were for practical application of the intervention. This was conducted with five CPR-B training torsos (Little Anne QCPR training mannequin, Laerdal) and a simulated AED for CPR training (AED Practi-Trainer - Bilingual, WNL). Both theoretical and practical training were provided by a basic life support instructor from the Spanish Society of Intensive Care Medicine and Coronary Units (SEMICYUC), instructing participants under the 2021 European Resuscitation Council (ERC) recommendations.
  Interventions: Other: PCR Trainning

INTERVENTIONS:
Other: PCR Trainning — A two-hour training intervention was conducted by a CPR-B instructor. The first 30 minutes were dedicated to explaining how to recognize a cardiopulmonary arrest, the correct technique for chest compressions, ventilations, and AED use. The remaining 90 minutes were for practical application of the intervention. This was conducted with five CPR-B training torsos (Little Anne QCPR training mannequin, Laerdal) and a simulated AED for CPR training (AED Practi-Trainer - Bilingual, WNL). Both theoretical and practical training were provided by a basic life support instructor from the Spanish Society of Intensive Care Medicine and Coronary Units (SEMICYUC), instructing participants under the 2021 European Resuscitation Council (ERC) recommendations.

SUMMARY:
This study aims to evaluate the change in attitudes and knowledge about basic cardiopulmonary resuscitation (CPR-B) in football professionals following a training intervention and to examine its correlation with sociodemographic variables.

The study consists of two phases. The first phase involves an observational cross-sectional study to assess the level of attitude and knowledge in cardiopulmonary resuscitation. The second phase includes an educational intervention consisting of a training and practical session on CPR-B, with a pre-post intra-subject control. The questionnaire was completed by football professionals from the Spanish first division and their coaches, with N=206 in the first phase and N=70 30 days after the training intervention in the second phase.

ELIGIBILITY:
Inclusion Criteria:

* being professional football players or coaches in the Valencian Community
* accept voluntarily participating in the study. All participants gave their written consent after being informed.

Exclusion Criteria:

* Not completing the questionnaire correctly (missing data)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in attitudes and knowledge about CPR-B | One month
  The goal is to evaluate the change in attitudes and knowledge about CPR-B in football professionals following a training intervention and to examine its correlation with sociodemographic variables. Validated questionnaires were used to assess the attitude towards helping others in CPR-B for both lay first responders and healthcare professionals(19) and those by Chein and Oteir to assess CPR-B knowledge(20-21). Additionally, some questions about CPR knowledge, based on the CPR knowledge questionnaire by Pivač and his team(19), were added and validated by an expert committee to check their relevance. The resulting questionnaire, comprising 48 items, was analyzed before and after the intervention, and statistical analysis was conducted on the sociodemographic variables (gender, education level, role of participants).

CONTACTS AND LOCATIONS:
Locations (1):
- Héctor Uso Vicent, Villarreal, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No
Professional soccer players are very well known and could jeopardize their career. The data belongs to the Football Club. On the other hand, upon request, we could share the encrypted database.

REFERENCES:
- See also: Related Info — https://www.erc.edu/